CLINICAL TRIAL: NCT01982422
Title: Developmental Origins of Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Joel Nigg, Ph.D., Director, Division of Psychology and Professor of Psychiatry, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6749
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Inattention; Impulsivity; Anxiety
Keywords: Attention Deficit and Hyperactivity Disorder; Nutrition; Diet; Developmental Origins of Disease
MeSH Terms: conditions — Impulsive Behavior; Anxiety Disorders; Attention Deficit Disorder with Hyperactivity; Developmental Origins of Health and Disease | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary Intervention (Experimental): A whole food, nutrient-dense dietary intervention which restricts processed foods high in food additives and optimizes micronutrient intake.
  Interventions: Behavioral: Whole Food, Nutrient-Dense Dietary Intervention
- Standard-of Care Group (Placebo Comparator): This group will receive normal standard-of-care for pregnancy.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Whole Food, Nutrient-Dense Dietary Intervention — The dietary intervention will be a whole food, nutrient-dense diet which restricts processed foods high in food additives while optimizing micronutrient intake.
  Arms: Dietary Intervention
Behavioral: Standard of Care — Normal standard-of-care for pregnancy.
  Arms: Standard-of Care Group

SUMMARY:
This is a study evaluating the relationship between prenatal nutrition and neural development in infants born to mothers with Attention Deficit Hyperactivity Disorder (ADHD). We are hypothesizing that women randomized to a whole food, nutrient-dense diet during their 3rd trimester of pregnancy will have infants with more advanced neural development as compared to infants born to mothers receiving standard-of-care treatment.

DETAILED DESCRIPTION:
Pregnant women with ADHD will be recruited from the patient population at Oregon Health & Science University (OHSU). They will be recruited during their 1st or 2nd trimester. After consent, baseline measures will be collected including height, weight, body composition measurements using calipers, 24-hour dietary recalls, and blood and urine samples. Women will also complete questionnaires regarding ADHD symptoms, stress, depression, and lifestyle. Women will be given a one-week food diary to fill out at home, which will be mailed in upon completion. Upon receipt of the food diary, women will be randomized into either a nutrition intervention group or a standard-of-care group. Women who are randomized to the intervention group will receive individual nutritional counseling every 2 weeks during their 3rd trimester of pregnancy. Before delivery, the baseline measures described above will again be collected. At delivery, placenta and cord blood samples will be taken. After birth, the infant will undergo an MRI between 2 and 5 weeks of age. The scan is completed while the baby sleeps, and special ear protection is worn to limit sleep disruption from the noise of the MRI. When the infant is 3 months old, mothers will complete questionnaires about infant feeding, sleep and behavior.

ELIGIBILITY:
Inclusion Criteria:

* Women in general good health
* 18 years of age or older
* Confirmed pregnancy and currently between 8 and 24 weeks pregnant
* With symptoms of inattention or impulsivity

Exclusion Criteria:

* Obstetrician confirmed high-risk pregnancy
* Current drug/alcohol addiction
* Current smoker
* Unwilling/unable to discontinue psychiatric medication during pregnancy
* Comorbid schizophrenia, bipolar, or major depressive disorder

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-08; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Functional neuroconnectivity of neonate assessed by MRI | 2-5 weeks after birth
  MRI will be used to examine brain morphology and functional connectivity in the neonates.

SECONDARY OUTCOMES:
Blood nutrient concentrations | Assessed at consent and end of 3rd trimester
  Maternal blood nutrient concentrations will be examined to assess whether or not the intervention group had higher nutrient levels in the 3rd trimester than the standard-of-care group.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Nigg, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States